CLINICAL TRIAL: NCT06705088
Title: A First-In-Human, Randomized, Double-Blind, Placebo-Controlled, Single And Multiple Ascending Oral Dose Study Of SUVN-I6107 To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics In Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics And Pharmacodynamics of SUVN-I6107 In Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: S1-I6107
Record Dates: First submitted 2024-11-14; First posted 2024-11-26 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: SUVN-I6107; First-in-Human; Muscarinic M1 Receptor Positive Allosteric Modulator (M1-PAM)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (Experimental): single ascending doses administered orally
  Interventions: Drug: SUVN-I6107; Drug: Placebo
- Multiple Ascending Dose (Experimental): multiple ascending doses administered orally for 14 days.
  Interventions: Drug: SUVN-I6107; Drug: Placebo

INTERVENTIONS:
Drug: SUVN-I6107 — SUVN-I6107 Tablet
Drug: Placebo — A look-alike tablet with no active ingredient.

SUMMARY:
The purpose of this study is 1) to investigate how safe and tolerable SUVN-I6107 is after a single oral dose at increasing dose levels and multiple oral doses at increasing dose levels, 2) to determine the pharmacokinetic (PK) profile after single and multiple ascending oral doses, 3) to investigate the effects of food on SUVN-I6107 pharmacokinetics and 4) to evaluate the pharmacodynamic (PD) effects of single and multiple ascending oral doses of SUVN-I6107 on quantitative electroencephalogram (qEEG) and event-related potential (ERP) assessments.

DETAILED DESCRIPTION:
This research study is a randomized, single-center, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD), first-in-human study in healthy participants.

This study consist of 2 segments: Segment 1 will be the SAD portion and Segment 2 will be the MAD portion.

Segment 1 will include up to 5 sequential cohorts. Up to 40 healthy male or female subjects, ages 18 - 45 years (inclusive) old at screening will be enrolled.

Segment 2 will include up to 3 sequential cohorts. The dosing will be administered for 14 consecutive days. Up to 24 healthy male or female subjects, ages 50 to 80 years (inclusive) old at screening will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): 18.0 to 30.0 kg/m2 for Segment 1 and 18.0 to 32.0 kg/m2 for Segment 2, inclusive, at screening and weight at least 50 kg and no more than 100 kg.
* Ability and willingness to abstain from alcohol-, caffeine-, and methylxanthine-containing beverages or food (eg, coffee, tea, cola, chocolate, energy drinks) from 48 hours (2 days) prior to each admission to the clinical facility until study discharge.
* All values for hematology and clinical chemistry tests of blood and urine within the normal range or showing no clinically relevant deviations, as judged by the Investigator, at screening and at admission.

Exclusion Criteria:

* Females who are pregnant, lactating, planning to become pregnant, or planning to donate ova/oocytes during this study or within 30 days after last administration of study drug.
* Males with female partners who are pregnant, lactating, or planning to become pregnant during this study or within 90 days after dosing of study drug.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of admission to the clinical site.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | From Day 1 to Day 11 (Segment 1) and from Day 1 to Day 24 (Segment 2)
  Number of participants with adverse events (AE), discontinuations due to AE or serious adverse event [SAE], and withdrawals from the study due to AE.
Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Values | From Baseline to Day 11 (Segment 1) and to Day 24 (Segment 2)
  Descriptive statistics of QTcF for observed values and changes from baseline will be summarized at each scheduled time point.
Number of Participants With Clinically Significant Changes in Blood Pressure | From baseline to Day 11 (Segment 1) and to Day 24 (Segment 2)
Number of Participants With Clinically Significant Changes in Pulse Rate | From baseline to Day 11 (Segment 1) and to Day 24 (Segment 2)
Number of Participants With Clinically Significant Changes in Body Temperature | From baseline to Day 11 (Segment 1) and to Day 24 (Segment 2)
Number of Participants With Clinically Significant Changes in Respiration Rate | From baseline to Day 11 (Segment 1) and to Day 24 (Segment 2)
Changes in Columbia Suicide Severity Rating Scale (C-SSRS) Score | From baseline to Day 24 (Segment 2)
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) | Day 1 and Day 14
  SUVN-I6107 concentrations levels will be assessed after single and multiple ascending oral doses.
Maximum observed concentration (Cmax) | Day 1 and Day 14
  SUVN-I6107 maximum observed concentration will be assessed after single and multiple ascending oral doses.
Time to reach maximum concentration (Tmax) | Day 1 and Day 14
  Time to reach maximum concentration will be assessed after single and multiple ascending oral doses.
Terminal half-life (t½) | Day 1 and Day 14
  SUVN-I6107 elimination rate will be assessed after single and multiple ascending oral doses.

OTHER OUTCOMES:
Quantitative electroencephalogram (qEEG) | Day 1 (Segment 1); Day 7 and Day 12 (Segment 2)
  Change in absolute quantitative electroencephalogram (qEEG) power from predose to postdose.
Latency for parameter from the Active, Auditory Oddball Event-related potential (ERP) test | Day 1 (Segment 1); Day 7 and Day 12 (Segment 2)
  Change in latency (in milliseconds) for the P300 parameter from the Active, Auditory Oddball ERP test from predose to postdose.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No